CLINICAL TRIAL: NCT05716464
Title: The Effect of Group-based Lifestyle Medicine Intervention and Cognitive Behavioural Therapy on Depressive Symptoms: A Pilot Randomised Controlled Trial
Brief Title: The Effect of Group-based Lifestyle Medicine Intervention and CBT on Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY029
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Depression
Keywords: Depression; Lifestyle medicine; Cognitive-behavioral therapy for depression; Randomised controlled trial
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle medicine intervention (LM) (Experimental): Participants in the LM group will receive a 6-week group-based lifestyle medicine intervention.
  Interventions: Behavioral: Lifestyle medicine intervention
- Cognitive-behavioral therapy for depression (CBT-D) (Experimental): Participants in the CBT-D group will receive a 6-week group-based cognitive-behavioral therapy for depression.
  Interventions: Behavioral: Cognitive-behavioral therapy for depression (CBT-D)

INTERVENTIONS:
Behavioral: Lifestyle medicine intervention — The lifestyle medicine intervention includes six weekly sessions (i.e., participants will receive the intervention once per week) that are related to the following topics: (a) lifestyle psychoeducation, (b) physical activity, (c) dietary recommendation, (d) stress management, (e) sleep management and (f) motivation and goal-setting techniques. Each topic will be delivered during each face-to-face session and the duration of each session will be around 120 minutes.
  Arms: Lifestyle medicine intervention (LM)
Behavioral: Cognitive-behavioral therapy for depression (CBT-D) — The group-based CBT-D therapy includes six weekly sessions (i.e., participants will attend one 120-minute, face-to-face group therapy per week, and will be asked to practice taught-skills every day, for 42 days) that are related to the following topics: (a) psychoeducation, (b) cognitive restructuring, (c) behavioral activation, (d) self-care and relapse prevention.
  Arms: Cognitive-behavioral therapy for depression (CBT-D)

SUMMARY:
The objective of this randomized controlled trial is to evaluate and compare the efficacy of group-based lifestyle medicine intervention and cognitive-behavioral therapy for depression (CBT-D) for Chinese adults with depressive symptoms.

Prior to all study procedures, eligible participants will be required to complete an online informed consent (with telephone support). Around 40 eligible participants aged between 18 to 65 with depression (Patient Health Questionnaire-9 [PHQ-9] ≥ 10) will be randomly assigned to the Lifestyle Medicine group (LM group), or the CBT-D group in a ratio of 1:1. Participants in both groups will receive interventions either through lifestyle medicine intervention or CBT-D group therapy for 6 consecutive weeks. The outcomes of interest will include depressive, anxiety, and insomnia symptoms, quality of life, functional impairment, and health-promoting behaviours at baseline (week 0), immediate (week 7) and 3-month post-intervention assessments (week 19). Treatment credibility and acceptability will be collected before and immediately after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults reside in Hong Kong;
2. Aged between 18 to 65 years;
3. Have a Patient Health Questionnaire-9 (PHQ-9) score ≥ 10, indicating at least moderate level of depressive symptoms;
4. Able to read and understand Chinese/Cantonese and are fluent in Cantonese;
5. Willing to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Received psychotherapy for depression in the past 6 months;
2. A change in psychotropic drugs that target depression within 2 weeks before the baseline assessment;
3. A PHQ-9 question 9 score higher than 2, indicating a moderate level of suicidal risk that requires active crisis management (referral information to professional mental health services will be provided);
4. Currently participating in another intervention study that may potentially improve mental health;
5. Self-disclosure of any psychiatric, medical or neurocognitive disorder(s) that makes participation unsuitable based on the team's clinical experience or interferes with adherence to the lifestyle modification (e.g., where exercise is not recommended by physicians);
6. Pregnancy;
7. Hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediate post-treatment, and 12-week follow-up
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediate post-treatment, and 12-week follow-up
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-treatment, and 12-week follow-up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediate post-treatment, and 12-week follow-up
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP-II) | Baseline, immediate post-treatment, and 12-week follow-up
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediate post-treatment, and 12-week follow-up
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success. Specific wording referencing "anxiety" was changed to refer to "depression".
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediate post-treatment, and 12-week follow-up
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from a short form of the International Physical Activity Questionnaire - Chinese version a short form of the IPAQ-C. The questions include: "On a typical weekday in the last 7 days, how many hours per day did you typically spend sitting?"; "On a typical weekend in the last 7 days, how many hours per day did you typically spend sitting?"; "During the last 7 days, on how many days did you do at least 10 minutes moderate physical activity/vigorous physical activity/walking?"; "How much time did you usually spend doing the moderate physical activity /vigorous physical activity/walking on one of those days?"; and "How much time did you usually spend engaging in physical activity while seated and standing on one of those days?"
Change in the Treatment Acceptability and Adherence Scale (TAAS) | Baseline and immediate post-treatment
  TAAS is a self-reported, ten-item questionnaire that is rated by a seven-point Likert scale from 1 to 7, and it aims at evaluating the clients' attitude toward the treatment sessions by four domains, including acceptability, adherence, drop-out, and distress. Specific wording referencing "anxiety" was changed to refer to "depression".

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Yan-Yee Ho, PhD, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No